CLINICAL TRIAL: NCT00361231
Title: Phase II Study of Gemcitabine, Oxaliplatin in Combination With Bevacizumab (Avastin) in Unresectable or Metastatic Biliary Tract and Gallbladder Cancer
Brief Title: Gemcitabine, Oxaliplatin in Combination With Bevacizumab in Biliary Tract and Gallbladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry); Sanofi (Industry); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Andrew X. Zhu, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-349
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Biliary Tract Cancer; Gallbladder Adenocarcinoma
Keywords: Avastin; GEMOX
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Bevacizumab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab, Gemcitabine, Oxaliplatin (Experimental): * The chemotherapy drugs are given twice every 28 days. This 28 day period is called a cycle of study treatment.
  * Bevacizumab will be administered by IV over 90 minutes on day 1 and day 15. Gemcitabine will be administered by IV over 1 hour and 40 minutes on days 1 and 15 of each cycle. Oxaliplatin will be administered by IV for 2 hours on days 1 and 15 of each cycle.
  * Participants will continue to receive cycles of study treatment as long as their disease does not progress and they are not experiencing any serious side effects.
  Interventions: Drug: Bevacizumab; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Bevacizumab — Given intravenously on days 1 and 15 of each 28-day cycle. Participants may continue to receive study treatment as lond as their disease does not progress and they do not experience any serious side effects.
  Other Names: Avastin
Drug: Gemcitabine — Given intravenously on days 1 and 15 of each 28-day cycle. Participants may continue to receive study treatment as lond as their disease does not progress and they do not experience any serious side effects.
  Other Names: Gemzar
Drug: Oxaliplatin — Given intravenously on days 1 and 15 of each 28-day cycle. Participants may continue to receive study treatment as lond as their disease does not progress and they do not experience any serious side effects.
  Other Names: Eloxatin

SUMMARY:
The purposes of this study are to test the safety of bevacizumab when given in combination with gemcitabine and oxaliplatin and to see what effects (good and bad) this combination has on patients with cancer of bile duct or gallbladder. Bevacizumab has been shown to slow or stop cell growth in tumors by decreasing the blood supply to the tumors.

DETAILED DESCRIPTION:
* The chemotherapy drugs are given twice every 28 days. This 28 day period is called a cycle of study treatment.
* Bevacizumab will be administered by IV over 90 minutes on day 1 and day 15. Gemcitabine will be administered by IV over 1 hour and 40 minutes on days 1 and 15 of each cycle. Oxaliplatin will be administered by IV for 2 hours on days 1 and 15 of each cycle.
* The following tests and procedures will be performed on day 1 and day 15 or each cycle: physical examination; medical history; blood work; and urine test. A PET scan will be repeated at the end of cycle 2 and CT scans will be repeated once every 8 weeks.
* Participants will continue to receive cycles of study treatment as long as their disease does not progress and they are not experiencing any serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally unresectable or metastatic biliary tract or gallbladder adenocarcinoma. Patients must have at least one measurable lesion outside prior radiation field.
* Zero to one prior chemotherapy for biliary tract or gallbladder cancer
* Age > 18 years
* ECOG performance status 0-2
* Life expectancy > 12 weeks
* Adequate organ and bone marrow function

Exclusion Criteria:

* Chemotherapy within past 3 weeks of initiation of therapy
* Pregnant or lactating women
* Clinically apparent central nervous system metastases or carcinomatous meningitis
* Biliary obstruction with inadequate drainage and total bilirubin > 2.5 mg/dL
* Concurrent malignancy of any site, except limited basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Uncontrolled serious medical or psychiatric illness
* Pre-existing peripheral neuropathy of grade 2 or greater severity according to the Common Terminology Criteria of the NCI (version 3.0)
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study
* Blood pressure of > 150/100 mmHg
* Unstable angina
* NYHA Grade II or greater congestive heart failure
* History of myocardial infarction or stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury with 28 days prior to Day 1, anticipation of need for major surgical procedure during the course of the study
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to day 1
* Serious, non-healing wound, ulcer, or bone fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-05; Primary Completion 2009-03 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew X. Zhu, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahani DV, Hayano K, Galluzzo A, Zhu AX. Measuring treatment response to systemic therapy and predicting outcome in biliary tract cancer: comparing tumor size, volume, density, and metabolism. AJR Am J Roentgenol. 2015 Apr;204(4):776-81. doi: 10.2214/AJR.14.13223. PMID 25794066
- [Derived] Zhu AX, Meyerhardt JA, Blaszkowsky LS, Kambadakone AR, Muzikansky A, Zheng H, Clark JW, Abrams TA, Chan JA, Enzinger PC, Bhargava P, Kwak EL, Allen JN, Jain SR, Stuart K, Horgan K, Sheehan S, Fuchs CS, Ryan DP, Sahani DV. Efficacy and safety of gemcitabine, oxaliplatin, and bevacizumab in advanced biliary-tract cancers and correlation of changes in 18-fluorodeoxyglucose PET with clinical outcome: a phase 2 study. Lancet Oncol. 2010 Jan;11(1):48-54. doi: 10.1016/S1470-2045(09)70333-X. Epub 2009 Nov 20. PMID 19932054

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab, Gemcitabine, Oxaliplatin: * The chemotherapy drugs are given twice every 28 days. This 28 day period is called a cycle of study treatment.
  * Bevacizumab will be administered by IV over 90 minutes on day 1 and day 15. Gemcitabine will be administered by IV over 1 hour and 40 minutes on days 1 and 15 of each cycle. Oxaliplatin will be administered by IV for 2 hours on days 1 and 15 of each cycle.
  * Participants will continue to receive cycles of study treatment as long as their disease does not progress and they are not experiencing any serious side effects.
  Bevacizumab: Given intravenously on days 1 and 15 of each 28-day cycle. Participants may continue to receive study treatment as lond as their disease does not progress and they do not experience any serious side effects.
  Gemcitabine: Given intravenously on days 1 and 15 of each 28-day cycle. Participants may continue to receive study treatment as lond as their disease does not progress and they do not experience any serious side effects.
Period: Overall Study
Arm/Group | Bevacizumab, Gemcitabine, Oxaliplatin
Started | 35
Completed | 1
Not Completed | 34
Not completed — Physician Decision | 3
Not completed — Symptomatic deterioration | 5
Not completed — Radiographic disease progression | 16
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 6

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab, Gemcitabine, Oxaliplatin
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 12
Age, Continuous [Median (Full Range); unit: years] | 60 [25 to 82]
Gender [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival
Description: To assess the median progression free survival in patients with BTC on GEMOX-B. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. In addition, death in the absence of radiological disease progression was also categorized as progression.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab, Gemcitabine, Oxaliplatin: * The chemotherapy drugs are given twice every 28 days. This 28 day period is called a cycle of studytreatment.
  * Bevacizumab will be administered by IV over 90 minutes on day 1 and day 15. Gemcitabine will be administered by IV over 1 hour and 40 minutes on days 1 and 15 of each cycle. Oxaliplatin will be administered by IV for 2 hours on days 1 and 15 of each cycle.
  * Participants will continue to receive cycles of study treatment as long as their disease does not progress and they are not experiencing any serious side effects.
  Bevacizumab: Given intravenously on days 1 and 15 of each 28-day cycle. Participants may continue to receive study treatment as lond as their disease does not progress and they do not experience any serious side effects.
  Gemcitabine: Given intravenously on days 1 and 15 of each 28-day cycle. Participants may continue to receive study treatment as lond as their disease does not progress and they do not experience any serious side effects.
  Oxaliplatin
Arm/Group | Bevacizumab, Gemcitabine, Oxaliplatin
Number analyzed (Participants) | 35
months | 7.0 [5.3 to 10.3]
Statistical Analysis 1: Comparison: Bevacizumab, Gemcitabine, Oxaliplatin; Test type: Superiority or Other; p < 0.05, Kaplan-Meier

2. Secondary Outcome: Overall Response Rate
Description: To assess the overall response rate of GEMOX-B in patients with advanced BTC. Response rate is determined through Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab, Gemcitabine, Oxaliplatin
Number analyzed (Participants) | 35
percentage of participants | 0
Statistical Analysis 1: Comparison: Bevacizumab, Gemcitabine, Oxaliplatin; Test type: Superiority or Other; p = 0.05, Kaplan-Meier

ADVERSE EVENTS:
Time Frame: May 17, 2006 and December 5, 2007
Groups:
- Bevacizumab, Gemcitabine, Oxaliplatin: * The chemotherapy drugs are given twice every 28 days. This 28 day period is called a cycle of study treatment.
  * Bevacizumab will be administered by IV over 90 minutes on day 1 and day 15. Gemcitabine will be administered by IV over 1 hour and 40 minutes on days 1 and 15 of each cycle. Oxaliplatin will be administered by IV for 2 hours on days 1 and 15 of each cycle.
  * Participants will continue to receive cycles of study treatment as long as their disease does not progress and they are not experiencing any serious side effects.
  Bevacizumab: Given intravenously on days 1 and 15 of each 28-day cycle. Participants may continue to receive study treatment as lond as their disease does not progress and they do not experience any serious side effects.
  Gemcitabine: Given intravenously on days 1 and 15 of each 28-day cycle. Participants may continue to receive study treatment as long as their disease does not progress and they do not experience any serious side eff
Arm/Group | Bevacizumab, Gemcitabine, Oxaliplatin
Serious Adverse Events (participants affected / at risk) | 12/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, Gemcitabine, Oxaliplatin (N=35)
Grade 4 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 — unlikely related
Grade 4 confusion (Nervous system disorders) | 2 — unrelated
Grade 3 Bilirubin (Investigations) | 1
Death within 30 days (General disorders) | 1 — Unrelated
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Grade 4 Cognitive disturbance (Nervous system disorders) | 1
Grade 4 Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Absolute Neutrophil Count (Blood and lymphatic system disorders) | 2 — Probably related
Grade 4 Hypophosphatemia (Metabolism and nutrition disorders) | 1 — (unlikely related)
Grade 4 lymphopenia (Blood and lymphatic system disorders) | 1 — probably related
Grade 4 fatigue (General disorders) | 2 — possibly related
Grade 3 Wound dehiscence (Blood and lymphatic system disorders) | 1
Grade 3 infection, wound (Infections and infestations) | 1
Grade 3 Hypoxia (General disorders) | 1
Grade 3 abdominal pain (Gastrointestinal disorders) | 1 — unrelated
Grade 4 Sepsis (Infections and infestations) | 1 — unlikely related
Acute myocardial infarction (Cardiac disorders) | 1 — possibly related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab, Gemcitabine, Oxaliplatin (N=35)
Leucopenia (Blood and lymphatic system disorders) | 24
Neutropenia (Blood and lymphatic system disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 26
Anaemia (Blood and lymphatic system disorders) | 26
Lymphopenia (Blood and lymphatic system disorders) | 15
Fatigue (General disorders) | 29
Neuropathy (Nervous system disorders) | 28
Raised AST (Gastrointestinal disorders) | 28
Nausea (Gastrointestinal disorders) | 27
Raised ALT (Gastrointestinal disorders) | 26
Constipation (Gastrointestinal disorders) | 21
Anorexia (Metabolism and nutrition disorders) | 20
Raised Alkaline phosphatase (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 14
Fever (General disorders) | 12
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11
Weight loss (Metabolism and nutrition disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Stomatitis (Gastrointestinal disorders) | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 7
Acne rash (Skin and subcutaneous tissue disorders) | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Allergic reaction (Immune system disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 5
Epistaxis (General disorders) | 16
Hypertension (Cardiac disorders) | 15
Headache (Nervous system disorders) | 13
Proteinuria (Metabolism and nutrition disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No